CLINICAL TRIAL: NCT05605782
Title: ORION (Ozanimod Real-World Safety - A Post- Authorisation Multi-National Long-term Non-Interventional Study)
Brief Title: A Post-Authorization, Long-term Study of Ozanimod Real-world Safety
Acronym: ORION
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-009; EUPAS44615 (Registry Identifier: EU PAS Registry)
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing-Remitting Multiple Sclerosis; Ozanimod; Serious opportunistic infections; Serious acute liver injury; Malignancy; Macular edema
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Neoplasms; Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Participants initiating treatment with ozanimod
- Participants initiating an sphingosine-1 phosphate (S1P) modulator
- Participants initiating other non-S1P-receptor modulators disease modifying treatments (DMTs)

SUMMARY:
The purpose of this study is to determine the rates of adverse events of interest (AEIs) in a real-world population of participants with relapsing remitting multiple sclerosis (RRMS) receiving Ozanimod, sphingosine-1 phosphate (S1P) receptor modulator, compared to the rates of these events in two population of participants:

* Participants not exposed to ozanimod with RRMS who have received treatment with other S1P-receptor modulators disease modifying treatments (DMTs)
* Participants not exposed to ozanimod with RRMS who have received treatment with other non-S1P-receptor modulators disease modifying treatments (DMTs)

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of multiple sclerosis (MS) recorded on or before the index prescription
* Have at least 6 months of continuous enrollment in the data source (thereby providing medical and dispensing/prescription history data, along with an operational definition of new use) before the index date

Exclusion Criteria:

• Participants with dispensing/prescription of more than one cohort defining drug on the index date

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include men and women at least 18 years old who have a diagnosis of multiple sclerosis and are new users of ("initiate") treatment with one of three cohort-defining treatments. Participants will be grouped into the following cohorts:
  * Exposed: Starting ozanimod
  * Non-exposed: Starting another sphingosine 1-phosphate (S1P) receptor modulator
  * Non-exposed: Starting a disease modifying treatment other than an S1P receptor modulator
Sampling Method: Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2033-07-26 (Estimated); Study Completion 2033-07-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular events (MACE) | Up to 10 years
Incidence of serious opportunistic infection (SOI) | Up to 10 years
Incidence of serious acute liver injury (SALI) | Up to 10 years
Incidence of macular edema | Up to 10 years
Identified rate of malignancies identified based upon the presence of at least 1 international classification of diseases, Tenth Revision, Clinical Modification (ICD-10-CM) diagnosis code | Up to approximately 2 years

SECONDARY OUTCOMES:
Incidence of symptomatic bradycardia | Up to approximately 5 years
Incidence of progressive multifocal leukoencephalopathy (PML) | Up to approximately 5 years
Incidence of posterior reversible encephalopathy syndrome (PRES) | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Evidera, Bethesda, Maryland, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html